CLINICAL TRIAL: NCT06121271
Title: Trial of Lu-177 DOTATATE (Lutathera®) in Unlicensed Indications Including Bronchial and Thymic Neuroendocrine Tumour, Paraganglioma/Phaeochromocytoma, Medullary Thyroid Carcinoma, and Repeat Peptide Receptor Radionuclide Therapy
Brief Title: Trial of Lu-177 DOTATATE (Lutathera®) in Unlicensed Indications
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 139005
Record Dates: First submitted 2022-02-08; First posted 2023-11-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Bronchial and Thymic Neuroendocrine Tumour; Paraganglioma/ Phaeochromocytoma; Medullary Thyroid Carcinoma; Those Requiring Repeat Peptide Receptor Radionuclide Therapy
MeSH Terms: conditions — Carcinoma, Medullary | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bronchial and Thymic Neuroendocrine Tumour (Experimental)
  Interventions: Drug: Lu-177 DOTATATE (Lutathera®)
- Paraganglioma/ Phaeochromocytoma (Experimental)
  Interventions: Drug: Lu-177 DOTATATE (Lutathera®)
- Medullary Thyroid Carcinoma (Experimental)
  Interventions: Drug: Lu-177 DOTATATE (Lutathera®)
- Those Requiring Repeat Peptide Receptor Radionuclide Therapy (Experimental)
  Interventions: Drug: Lu-177 DOTATATE (Lutathera®)

INTERVENTIONS:
Drug: Lu-177 DOTATATE (Lutathera®) — Treatment with Lutathera will consist of a total cumulative intravenous (IV) administered radioactivity dose of 29.6 GBq (800 mCi) or 14.8 GBq (400 mCi) for 4 cycles or 2 cycles of Lutathera, respectively.

SUMMARY:
This study is a phase 2, open, single-site trial. The primary objective of this study is to prospectively evaluate the safety and efficacy in participants treated with Lu-177 DOTATATE (Lutathera) in unresectable or metastatic, somatostatin receptor-expressing neuroendocrine tumours (NET) in currently unlicensed indications (eg, bronchial and thymic NET; paraganglioma/phaeochromocytoma; medullary thyroid carcinoma; and those requiring repeat peptide receptor radionuclide therapy (PRRT) with 2 further cycles of Lutathera). The aim is to recruit a total of 75-110 participants. Each patient will receive 4 cycles of Lutathera with 8-12 weeks time interval (except patients requiring repeat PRRT will receive 2 further cycles of Lutathera). The follow-up period will be for 2 years from the date of the last treatment.

DETAILED DESCRIPTION:
This clinical study is being conducted at the Royal Free Hospital / London. A total of 75-110 participants will be enrolled based on multidisciplinary team decisions and after meeting the criteria for enrollment.

Patients involved will be classified into the following subgroups:

Repeat PRRT if the participant have had the PRRT treatment before (2 cycles each): 35-45 participants Bronchial NET (4 cycles each): 25-35 participants Paraganglioma or phaeochromocytopma (4 cycles each): 10-20 participants Others NETs (eg, MedullaryThyroid Carcinoma) (4 cycles each): 5-10 participants The duration of study participation for all patients will be 24 months. After the participant signed the Informed Consent Form, he/she will be asked to undergo several screening investigations and procedures to ensure they are appropriate for the treatment and study. The screening takes place between 90 days and 1 day before treatment. Screening evaluations will include a review of the previous scans and blood tests. It is possible that in this period the participant might need an additional scan or blood test to ensure the participant meets the requirements of the study. During visits, the research doctor or nurse will take a relevant medical history and perform a physical exam and check the vital signs. The participant will be asked to fill a Quality-of-Life questionnaire.

Then blood and urine samples will be taken from the participant and will be sent to the laboratory for analysis. The participant will also be sent for a scan to assess heart function.

Treatment Phase:

Therapy Visits (Week 0,8,16,24):

The participant will be interviewed by the research doctor /nurse and will be asked few questions related to cancer and general health. A blood sample will be taken and sent for analysis. The radiopeptide 177Lu-DOTATATE will be administered as a slow intravenous infusion via a cannula into a vein in the arm. The infusion will last 20 to 30 minutes. In addition to the 177Lu-DOTATATE administration, the participant will receive an amino acid solution (AAS) which is given to protect kidneys from radiation. The amino acid solution is infused over 4 - 6 hours, starting 30 - 60 minutes before PRRT via the same cannula.

After infusion of 177Lu-DOTATATE, the participant's vital signs (temperature, pulse and blood pressure) will be checked.

Around 4 hours after each therapy administration the participant will have imaging with a scan in the nuclear medicine department to show that the tumour has taken up the treatment as expected. After 177Lu-DOTATATE the participant will receive a patient card with safety precautions to be taken after being administered the radioactive therapy. Post Therapy Visits (Week 4,12,20,28, and week 36) (performed at local GP or nurse at home).

A blood test will be taken to check that blood cells are in an appropriate range and that kidney function is at the recommended levels.

Follow-Up phase:

After completion of the 24 months, the participant will return to that usual protocol of CT or MRI scans every 6 months.

The participant will meet the study doctor/nurse as usual who will perform an examination and arrange the standard blood tests. The trial will be finished after 2 years from the date of the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age.
2. Participants capable of giving informed consent
3. Presence of unresectable or metastatic, well differentiated, somatostatin receptor positive non gastroenteropancreatic neuroendocrine tumours. Or for those having 2 cycles repeat therapy, GEP NET > 18 months from start of previous PRRT.
4. Patients must have progressive disease based on RECIST Criteria, Version 1.1. In order to make the assessment, two CT (or MRI) scans are required. The oldest scan must not be older than 3 years from the date of enrolment. The most recent scan must not be older than 6 weeks from the date of enrolment.
5. Confirmed presence of somatostatin receptors on all target lesions (for target/non-target/measurable lesions definition see RECIST Criteria, Version 1.1) documented by CT/MRI scans, based on positive OctreoScan or Ga68 Dotatate PET imaging within 24 weeks prior to enrolment in the trial.
6. The tumour uptake observed in each target lesion (for target/non-target/measurable lesions definition see RECIST Criteria, Version 1.1) using OctreoScan/Tc-99m-SRS should be ≥ normal liver uptake observed on planar imaging.
7. The tumour uptake observed in each target lesion (for target/non-target/ measurable lesions definition see RECIST Criteria, Version 1.1) using Ga68 Dotatate PET should be ≥ normal liver uptake observed on PET imaging.
8. KPS ≥60.
9. Presence of at least 1 measurable site of disease on cross-sectional imaging.
10. Females of childbearing potential (defined as <2 years after last menstruation and not surgically sterile) and males, who are not surgically sterile or with female partners of childbearing potential must be willing to use a highly effective method of contraception during treatment and for a minimum of 6 months after the end of treatment (hormonal or barrier method of birth control; abstinence). Contraceptive methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods. Such methods include:

    • combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:
    * oral
    * intravaginal
    * transdermal

      * progestogen-only hormonal contraception associated with inhibition of ovulation
    * oral
    * injectable
    * implantable

      • intrauterine device (IUD)

      • intrauterine hormone-releasing system (IUS)

      • bilateral tubal occlusion

      • vasectomised partner

      • sexual abstinence
      * Women of childbearing potential (WOCBP) must have a negative pregnancy test within 7 days prior to treatment initiation). NOTE: Participants are considered not of childbearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or they are postmenopausal. Inclusion Criteria for Subsequent Treatments

1. Both serum creatinine ≤150 μmol/L (≤1.7 mg/dL) and calculated creatinine clearance ≥40 mL/min, eventually confirmed by measured creatinine clearance (or measured GFR) using isotopic GFR measurement ≥40 mL/min (the measured creatinine clearance/GFR is required only as confirmatory exam).

2. Haemoglobin concentration ≥5.0 mmol/L (≥8.0 g/dL); WBC ≥2 x109/L (≥2000/mm3); platelets ≥75 x109/L (≥75 x103/mm3).

3. Total bilirubin ≤3x ULN. 4. Serum albumin >3.0 g/dL, or serum albumin ≤3.0 g/dL, but normal prothrombin time.

5. KPS ≥60.

Exclusion Criteria:

* Participants will not be eligible for trial participation if they meet any of the exclusion criteria, or will be discontinued at the discretion of the Investigator if they develop any of the exclusion criteria during the trial.

Exclusion Criteria at Baseline

1. Either serum creatinine >150 μmol/L (>1.7 mg/dL), or calculated creatinine clearance <40 mL/min, eventually confirmed by measured creatinine clearance (or measured GFR using isotopic GFR measurement) <40 mL/min (the measured creatinine clearance/GFR is required only as confirmatory exam).
2. Haemoglobin concentration <5.0 mmol/L (<8.0 g/dL); WBC <2 x109/L (2000/mm3); platelets <75 x109/L (75 x103/mm3).
3. Total bilirubin >3x upper limit of normal (ULN).
4. Serum albumin <3.0 g/dL unless prothrombin time is within the normal range.
5. Pregnancy, planning a pregnancy or lactation.
6. Any surgery, radioembolization, chemoembolization, chemotherapy, and radiofrequency ablation within 12 weeks prior to enrolment in the trial.
7. Interferon, Everolimus (mTOR-inhibitors), or other systemic therapies within 4 weeks prior to enrolment in the trial.
8. Patients with a history of brain metastases must have a head CT with contrast to document stable disease prior to enrolment in the trial.
9. Uncontrolled congestive heart failure (NYHA II, III, IV).
10. Uncontrolled diabetes mellitus as defined by a fasting blood glucose >2x ULN.
11. Any participant receiving treatment with short-acting Octreotide, which cannot be interrupted for 12 hours before and 24 hours after the administration of Lutathera, or any participant receiving treatment with Octreotide LAR or Lanreotide Autogel, which cannot be interrupted for at least 28 days before the administration of Lutathera, unless the tumour uptake observed on target and non-target but measurable lesions by OctreoScan or Ga68 Dotatate PET imaging during continued Octreotide LAR or Lanreotide Autogel treatment is at least as high as normal liver uptake observed by planar imaging (Kwekkeboom, Krenning et al. 2009).
12. Patients with any other significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with completion of the trial.
13. Prior external beam radiation therapy to more than 25% of the bone marrow.
14. Current spontaneous urinary incontinence.
15. Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and proven no evidence of recurrence for 5 years.
16. Patients who have not provided a signed ICF to participate in the trial, obtained prior to the start of any protocol related activities.
17. Patient with known incompatibility to CT Scans with IV contrast due to allergic reaction or renal insufficiency. If such participants can be imaged without the use of CT contrast material (ie, can tolerate MRI scans), such participants would not be excluded.
18. Patients who have participated in any therapeutic clinical trial/received any investigational agent within the last 30 days are excluded from participation in this trial.
19. Patients with hypersensitivity to Lutathera (active substance or any of the excipients).
20. Involved in the planning or conduct of this trial.
21. Unwilling or unlikely to comply with the requirements of the trial. Exclusion Criteria for Subsequent Treatments

1. Exclusion criteria for Baseline # 1, 2, 3, 4, and 10 apply to all subsequent treatments, when a relationship cannot be excluded with either trial drugs or the corresponding toxicity has not resolved.

2. In relation to renal function, participants are also excluded from further therapy in case of >40% increase of serum creatinine over the baseline and with a concomitant decrease of >40% in creatinine clearance as calculated according to the Cockroft-Gault method, eventually confirmed by measured creatinine clearance (or GFR), if a relationship may not be excluded and the corresponding toxicity has not resolved.

3. When such exclusion criteria events occur, the participant will postpone any subsequent trial treatment until resolution of the event (normalisation or return to baseline values). The participant remains in the trial and continues observation with the scheduled tumour and clinical assessments.

4. All other exclusion criteria for enrolment eligibility apply to all subsequent treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-12-18 (Estimated); Primary Completion 2027-11-06 (Estimated); Study Completion 2027-11-06 (Estimated)

PRIMARY OUTCOMES:
To prospectively evaluate safety in participants treated with Lu-177 DOTATATE (Lutathera) in somatostatin receptor-expressing neuroendocrine tumours (NET) in currently unlicensed indications | 4 years
  Treatment-related toxicity will be assessed in all participants by Common Terminology Criteria for Adverse Events [CTCAE] v5.0. This will be done by performing electrocardiograms (ECGs), vital signs, and clinical laboratory tests (haematology, clinical chemistry, or urinalysis)at the baseline and before and after every treatment and during the follow-up period.
To prospectively evaluate tolerability in participants treated with Lu-177 DOTATATE (Lutathera) in somatostatin receptor-expressing neuroendocrine tumours (NET) in currently unlicensed indications | 4 years
  Treatment-related side effects and cancer-related symptoms will be assessed in all participants Questionnaire after every treatment and during the follow-up period.
To prospectively evaluate efficacy in participants treated with Lu-177 DOTATATE (Lutathera) in somatostatin receptor expressing neuroendocrine tumours (NET) in currently unlicensed indications | 4 years
  The efficacy of Lu-177 DOTATATE is assessed in all participants by measuring Progression Free Survival (PFS) and defined as the time from the date of start of treatment the date of the first documented tumour progression or death due to any cause.

SECONDARY OUTCOMES:
• To determine the Objective Response Rate (ORR) | 2 years
  ORR is defined by evaluating post-therapy scans (using RECIST Criteria, Version 1.1) looking for the percentage of patients who had a partial response or complete response from the whole cohort over the treatment time of 2 years.
• To determine the Overall Survival (OS). | 4 years
  Overall Survival (OS) is defined as the time from the date of start of treatment till death or loss of contact or end of trial.

IPD SHARING:
Plan to Share IPD: No